CLINICAL TRIAL: NCT02043197
Title: Post-Marketing Observational Program of Fevarin® Effectiveness in Treatment of Depression in Patients With Neurological Disorders (FRIENDS)
Brief Title: Fevarin® Effectiveness in Treatment of Depression in Patients With Neurological Disorder
Acronym: FRIENDS
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: Manipal Acunova Ltd. (Network)
Responsible Party: Sponsor
Other Study IDs: P14-326
Record Dates: First submitted 2013-12-23; First posted 2014-01-23 (Estimated); Results first posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-06

CONDITIONS: Depression
Keywords: Depression,; depressive symptoms,; major depressive disorder,; Fevarine,; fluvoxamine,; cognitive function,; neurological disorders,; sleep state
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Outpatients with neurological disorders and depression.: Outpatients with mild or moderate symptoms of depression prescribed by Fevarin® in accordance with the approved local label.

SUMMARY:
Prospective, multicenter, non-comparative, observational program to describe prevalence of depressive symptoms in a variety of neurological disorders and effects of Fevarin® on the severity of anxiety and depression, sleep state, and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with neurological disorders and mild or moderate symptoms of depression with Hospital Anxiety Depression Scale (HADS) depression scale score of 8 and higher. Fevarin® prescribed not earlier than 7 days before Visit 1.

Exclusion Criteria:

* Labeled contraindications to Fevarin®, psychotic symptoms and/or suicidal ideation, schizophrenia, bipolar disorder, schizoaffective disorder, severe dementia, alcohol or drug abuse, acute neurological disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinics
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Vladimirova, MD, PhD, Study Director — Abbott
Locations (29):
- Russia (29):
  - Research Facility ID ORG-000890, Chelyabinsk
  - Research facility ID ORG-000881, Krasnoyarsk
  - Research facility ID ORG-000893, Moscow
  - Research facility ID ORG-000882, Moscow
  - Research facility ID ORG-000876, Moscow
  - Research facility ID ORG-000877, Moscow
  - Research Facility ID ORG-000889, Nizhny Novgorod
  - Research facility ID ORG-000880, Novosibirsk
  - Research Facility ID ORG-000879, Penza
  - Research facility ID ORG-000891, Perm
  - Research facility ID ORG-000840, Perm
  - Research facility ID ORG-000803, Rostov-on-Don
  - Research facility ID ORG-000898, Rostov-on-Don
  - Research facility ID ORG-001028, Rostov-on-Don
  - Research facility ID ORG-001027, Rostov-on-Don
  - Research facility ID ORG-000894, Rostov-on-Don
  - Research facility ID ORG-000896, Saint Petersburg
  - Research facility ID ORG-000892, Saint Petersburg
  - Research facility ID ORG-000965, Saint Petersburg
  - Research facility ID ORG-000897, Samara
  - Research facility ID ORG-000839, Saratov
  - Research Facility ID ORG-000873, Spassk-Dal'niy
  - Research Facility ID ORG-000878, Tver'
  - Research facility ID ORG-001026, Vladivostok
  - Research Facility ID ORG-000874, Volgograd
  - Research Facility ID ORG-000888, Volgograd
  - Research Facility ID ORG-000895, Voronezh
  - Research facilility ID ORG-000872, Yekaterinburg
  - Research facility ID ORG-000875, Yessentuki

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Outpatients With Neurological Disorders and Depression.
Started | 300
Completed | 292
Not Completed | 8

BASELINE CHARACTERISTICS:
Population: 299 patients were in the Intent-to-treat population 296 patients were in the Per Protocol population At each mesurement an actual number of assessed patients is presented
Arm/Group | Outpatients With Neurological Disorders and Depression.
Number analyzed (Participants) | 299
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 245
  >=65 years | 54
Age, Continuous [Mean (Full Range); unit: years] | 50.51 [21 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 219
  Male | 80
Region of Enrollment [Number; unit: participants]
  Russian Federation | 299

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Different Neurological Disorders Associated With Depression Treated With Fluvoxamine (Fevarin®).
Description: The primary neurologic diagnosis was coded according to International Classification of Diseases and Related Health Problems, revision 10 http://apps.who.int/classifications/icd10/browse/2010/en In the report all diseases were summarized by Classes. Percentage of patients reporting at least once a specified symptom during the treatment period.
Time Frame: Baseline
Population: The actual number of assessed patients was provided to each measure.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Outpatients With Neurological Disorders and Depression.
Number analyzed (Participants) | 299
Percentage
  International Classification of Diseases G00-G99 | 49.2 [43.4 to 55]
  International Classification of Diseases I00-I99 | 31.8 [26.5 to 37.4]
  International Classification of Diseases M00-M99 | 20.1 [15.7 to 25.1]
  International Classification of Diseases T00-T99 | 2.7 [1.2 to 5.2]

2. Secondary Outcome: Change in the Hospital Anxiety and Depression Scale (HADS) Depression Subscale Score
Description: HADS scale used under license agreement https://www.gl-assessment.co.uk/products/hospital-anxiety-and-depression-scale-hads/
  The scale have two subscales:
  HADS-Anxiety HADS-Depression
  Each subscale has range 0-21 with following interpretation:
  0-7 normal 8-10 mild 11-14 moderate 15-21 severe
  In this place 'Change in the Hospital Anxiety and Depression Scale (HADS) Depression Subscale Score' is presented
Time Frame: From Baseline up to Day 30 and Day 90
Population: The actual number of assessed patients was provided to each measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Outpatients With Neurological Disorders and Depression.
Number analyzed (Participants) | 296
units on a scale
  Baseline Day 30 | -3 (2.5)
  Baseline Day 90 | -6 (3.24)

3. Secondary Outcome: Percent of Patients With Change of Depression Symptoms From Baseline to Day 30
Time Frame: From Baseline up to Day 30
Population: The actual number of assessed patients was provided to each measure.
Measure: Number; unit: percentage of participants
Arm/Group | Outpatients With Neurological Disorders and Depression.
Number analyzed (Participants) | 296
percentage of participants
  Improved | 88.2
  Worsened | 2.7
  No change | 9.1

4. Secondary Outcome: Change in the Hospital Anxiety and Depression Scale (HADS) Anxiety Subscale Score
Description: HADS scale used under license agreement https://www.gl-assessment.co.uk/products/hospital-anxiety-and-depression-scale-hads/
  The scale have two subscales:
  HADS-Anxiety HADS-Depression
  Each subscale has range 0-21 with following interpretation:
  0-7 normal 8-10 mild 11-14 moderate 15-21 severe
  In this place 'Change in the Hospital Anxiety and Depression Scale (HADS) Anxiety Subscale Score' is presented
Time Frame: From Baseline up to Day 30 and Day 90
Population: The actual number of assessed patients was provided to each measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Outpatients With Neurological Disorders and Depression.
Number analyzed (Participants) | 296
units on a scale
  Baseline Day 30 | -3.4 (2.78)
  Baseline Day 90 | -6.5 (3.62)

5. Secondary Outcome: Change in the Clinical Condition Measured by Clinical Global Impression Scale - Severity of Illness Subscale
Description: Clinical Global Impression Scale (CGI) was used. CGI is in the public domain. Severity of illness is the subscale of Clinical Global Impression (CGI). Severity of illness - reported in this place 0 = Not assessed, 1 = Normal, not at all ill, 2 = Borderline mentally ill, 3 = Mildly ill, 4 = Moderately ill, 5 = Markedly ill, 6 = Severely ill, 7 = Among the most extremely ill patients
Time Frame: Baseline, Day 90
Population: The actual number of assessed patients was provided to each measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Outpatients With Neurological Disorders and Depression.
Number analyzed (Participants) | 288
units on a scale | -1 (0.91)

6. Secondary Outcome: Percent of Patients With Change in Clinical Global Impression Scale
Time Frame: From Baseline up to Day 90
Population: The actual number of assessed patients was provided to each measure.
Measure: Number; unit: percentage of participants
Arm/Group | Outpatients With Neurological Disorders and Depression.
Number analyzed (Participants) | 294
percentage of participants
  Very much improved | 38.1
  Much improved | 46.9
  Minimaly improved | 11.2
  No change | 2.4
  Minimaly worse | 0.3
  Much worse | 0.3
  Not assessed | 0.7

7. Secondary Outcome: Anxiety and Depression Symptoms Score Measured by Hospital Anxiety and Depression Scale (HADS)
Description: HADS scale used under license agreement https://www.gl-assessment.co.uk/products/hospital-anxiety-and-depression-scale-hads/
  The scale have two subscales:
  HADS-Anxiety HADS-Depression
  Each subscale has range 0-21 with following interpretation:
  0-7 normal 8-10 mild 11-14 moderate 15-21 severe
  In this place Change in the Hospital Anxiety and Depression Scale (HADS) Both Subscale Scores are presented assessed at Day 180
Time Frame: Up to 180 days
Population: The actual number of assessed patients was provided to each measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Outpatients With Neurological Disorders and Depression.
Number analyzed (Participants) | 239
units on a scale
  HADS - D | 4.2 (3.17)
  HADS - A | 4.7 (3.33)

8. Secondary Outcome: Percent of Patients With Change of Anxiety Symptoms From Baseline to Day 30.
Time Frame: From Baseline up to Day 30
Population: The actual number of assessed patients was provided to each measure.
Measure: Number; unit: percentage of participants
Arm/Group | Outpatients With Neurological Disorders and Depression.
Number analyzed (Participants) | 296
percentage of participants
  Improved | 89.9
  Worsened | 2.7
  No change | 7.4

9. Secondary Outcome: Gender
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Outpatients With Neurological Disorders and Depression.
Number analyzed (Participants) | 299
percentage of participants
  Female | 73.24
  Male | 26.76

10. Secondary Outcome: Race
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Outpatients With Neurological Disorders and Depression.
Number analyzed (Participants) | 299
percentage of participants
  Asian | 0.7
  White | 99.3

11. Secondary Outcome: Family Status
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Outpatients With Neurological Disorders and Depression.
Number analyzed (Participants) | 299
percentage of participants
  Civil marriage | 1
  Divorced | 5.4
  Married | 65.9
  Single | 15.7
  Widow(er) | 12

12. Secondary Outcome: Education
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Outpatients With Neurological Disorders and Depression.
Number analyzed (Participants) | 299
percentage of participants
  Elementary | 3
  Secondary | 33.8
  University | 63.2

13. Secondary Outcome: Employment
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Outpatients With Neurological Disorders and Depression.
Number analyzed (Participants) | 299
percentage of participants
  Employed | 62.5
  Unemployed | 37.5

14. Other Pre Specified Outcome: Cognitive Functions Measured by Montreal Cognitive Assessment (MOCA)
Description: MoCA test used under license agreement www.mocatest.org
  Scale range 0-30 Normal >=26 Higher values represent a better outcome
Time Frame: Baseline, Day 90, Up to 180 days
Population: The actual number of assessed patients was provided to each measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Outpatients With Neurological Disorders and Depression.
Number analyzed (Participants) | 296
units on a scale
  Baseline | 25.2 (3.63)
  Day 90 | 27 (2.69)
  Day 180 | 27.5 (2.42)

15. Other Pre Specified Outcome: Insomnia Severity Index
Description: Insomnia Severity Index (ISI) used under license agreement cmorin@psy.ulaval.ca
  Total score has the range from 0 to 28 points with the following categories:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe). Higher values represent a worse outcome
Time Frame: Baseline, Day 90, Up to 180 days
Population: The actual number of assessed patients was provided to each measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Outpatients With Neurological Disorders and Depression.
Number analyzed (Participants) | 296
units on a scale
  Baseline | 13.4 (5.52)
  Day 90 | 6.6 (4.32)
  Day 180 | 4.5 (3.98)

16. Other Pre Specified Outcome: Percent of Patients With Quality of Sleep Change Assessed by Insomnia Severity Index (ISI) at Day 90
Description: Percent of Patients With Quality of Sleep Change Assessed by Insomnia Severity Index (ISI) From Baseline to Day 90.
Time Frame: From baseline up to Day 90
Population: The actual number of assessed patients was provided to each measure.
Measure: Number; unit: percentage of participants
Arm/Group | Outpatients With Neurological Disorders and Depression.
Number analyzed (Participants) | 294
percentage of participants
  Improved | 91.5
  Worsened | 4.1
  No change | 4.4

17. Other Pre Specified Outcome: Change in the Clinical Condition Measured by Clinical Global Impression Scale - Severity of Illness Subscale From Day 90 to 180 Days
Description: as for outcome 5
Time Frame: From Day 90 up to Up to 180 days
Population: The actual number of assessed patients was provided to each measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Outpatients With Neurological Disorders and Depression.
Number analyzed (Participants) | 239
units on a scale | -0.2 (0.55)

18. Other Pre Specified Outcome: Percent of Patients With Change in Clinical Global Impression Scale - Global Improvement Subscale Assessed at Day 180
Description: Global improvement - qualitative scale 0 = Not assessed, 1 = Very much improved , 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse
Time Frame: From Day 90 up to 180 days
Population: The actual number of assessed patients was provided to each measure.
Measure: Number; unit: percentage of participants
Arm/Group | Outpatients With Neurological Disorders and Depression.
Number analyzed (Participants) | 298
percentage of participants
  Very much improved | 56.9
  Much improved | 29.3
  Minimaly improved | 9.6
  No change | 2.9
  Minimaly worse | 0.8
  Much worse | 0.4

ADVERSE EVENTS:
Description: 299 patients were in the Intent-to-treat population
Arm/Group | Outpatients With Neurological Disorders and Depression.
All-Cause Mortality (participants affected / at risk) | 0/299
Serious Adverse Events (participants affected / at risk) | 0/299
Other Adverse Events (participants affected / at risk) | 22/299
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Outpatients With Neurological Disorders and Depression. (N=299)
Palpitations (Cardiac disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Asthenia (General disorders) | 5 (5)
Drug ineffective (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Coordination abnormal (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 3 (3)
Hyperkinesia (Nervous system disorders) | 1 (1)
Postural tremor (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 4 (4)
Tremor (Nervous system disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 2 (2)
Psychogenic tremor (Psychiatric disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No